CLINICAL TRIAL: NCT01467648
Title: The Pharmacodynamics of Doripenem Between 4-hour and 1-hour Infusion in Patients With Ventilator-associated Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sutep Jaruratanasirikul (Other)
Collaborators: Prince of Songkla University (Other)
Responsible Party: Sponsor-Investigator, Sutep Jaruratanasirikul, Principal Investigator, Prince of Songkla University
Organization: Prince of Songkla University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DORINOS4004
Record Dates: First submitted 2011-10-31; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Ventilator-Associated Pneumonia
Keywords: Infection; Doripenem; Ventilator-Associated Pneumonia; pharmacokinetic; pharmacodynamic
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Infections | interventions — Doripenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5 g by 4 hour infusion (Experimental): Blood samples (approximately 2 ml) in group " 0.5 g of doripenem with 4 h infusion every 8 h regimen" will be obtained by direct venepuncture at the following time: 0, 0.5, 1, 2, 3, 4, 4.5, 5, 6, 7 and 8 h after 7th dose of doripenem.
  Interventions: Drug: Doripenem
- 0.5 g by 1 hour infusion (Experimental): Blood samples (approximately 2 ml) in group " 0.5 g of doripenem with 1 h infusion every 8 h regimen" will be obtained by direct venepuncture at the following time: 1, 1.5, 2, 4, 5, 6, 7 and 8 h after 7th dose of doripenem.
  Interventions: Drug: Doripenem

INTERVENTIONS:
Drug: Doripenem — (i) 0.5 g in 100 ml of normal saline solution and administered via an infusion pump at a constant flow rate over 1 h every 8 h.
  Blood samples (approximately 2 ml)will be obtained by direct venepuncture at the following time: 0, 0.5, 1, 2, 3, 4, 4.5, 5, 6, 7 and 8 h after 7th dose of doripenem.
  Other Names: Doripenem (Doribax)
  Arms: 0.5 g by 4 hour infusion
Drug: Doripenem — (ii) 0.5 g in 100 ml of normal saline solution and administered via an infusion pump at a constant flow rate over 1 h every 8 h.
  Blood samples (approximately 2 ml) will be obtained by direct venepuncture at the following time: 1, 1.5, 2, 4, 5, 6, 7 and 8 h after 7th dose of doripenem.
  Other Names: Doripenem (Doribax)
  Arms: 0.5 g by 1 hour infusion

SUMMARY:
This is prospective and randomized study to assess the pharmacodynamics (t>MIC) of 0.5 g every 8 h of doripenem in patients with VAP following administration by a 4 h infusion or 1 h infusion.

Clinical and laboratory data such as Age,Sex, Body weight, Electrolyte, Vital signs, APACHE II score, BUN, Cr, Blood culture will be collected.

Twelve patients will be enrolled in this study. After completion of the doripenem therapy for 3 days in this study, all patients will receive other sensitive antibiotics to eradicate their bacterial infections.

Doripenem pharmacokinetic study will be carried out during the doripenem therapy. Blood samples (approximately 2 ml) in group " 0.5 g of doripenem with 4 h infusion every 8 h regimen" will be obtained by direct venepuncture at the following time: 0, 0.5, 1, 2, 3, 4, 4.5, 5, 6, 7 and 8 h after 7th dose of doripenem.

Blood samples (approximately 2 ml) in group " 0.5 g of doripenem with 1 h infusion every 8 h regimen" will be obtained by direct venepuncture at the following time: 1, 1.5, 2, 4, 5, 6, 7 and 8 h after 7th dose of doripenem.

The doripenem assays by method of Ikeda K et al. (J Chromatogr B, 2008) will be performed.

Concentration of doripenem in plasma will be simulated in Monte Carlo technique (Computer model) to get PK/PD index (40%T>MIC) and reported to % PTA (Probability Target Attainment) and %CFR (Cumulative Faction Response)

DETAILED DESCRIPTION:
Introduction:

The treatment of resistant pathogens is becoming more difficult, and only a few novel antimicrobial agents are currently in development with activity against highly resistant Gram negative bacteria. Doripenem is a carbapenem antibacterial agent with a broad spectrum of activity against Gram-negative and Gram-positive bacteria. This agent is often used as the last line of therapy for highly resistant Gram negative bacilli nosocomial pathogens. In common with other beta-lactam, the main pharmacokinetic/pharmacodynamic (PK/PD) index that correlates with the therapeutic efficacy is the time that concentrations in the tissue and serum are above the MIC (t>MIC). However, in tropical countries the stability of carbapenem antibiotics is an important consideration when considering continuous infusion. Therefore, prolonged infusion may be a useful route of administration to maximize bactericidal activity. In addition, pharmacokinetic changes have been found for several antimicrobial agents in critically ill patients, including ventilator-associated pneumonia. However, until now we have had no data to reveal the PK/PD index of doripenem in these critically ill patients.

Objectives:

To assess the pharmacodynamics (t>MIC) of 0.5 g every 8 h of doripenem in patients with VAP following administration by a 4 h infusion or 1 h infusion.

Clinical and laboratory data: Age,Sex, Body weight, Electrolyte, Vital signs, APACHE II score, BUN, Cr, Blood culture

Drug preparation and administration:

Doripenem will be reconstituted with saline solution according to the manufacturer's guidelines and then administered to the patients by 2 regimens:

1.0.5 g in 100 ml of normal saline solution and administered via an infusion pump at a constant flow rate over 4 h every 8 h.

2.0.5 g in 100 ml of normal saline solution and administered via an infusion pump at a constant flow rate over 1 h every 8 h.

Study design:

The study is planned as a prospective and randomized in patients with VAP. Each patients will receive doripenem in 2 regimens at room temperature (37°C) consecutively: (i) infusion of 0.5 g of doripenem for 4 h via an infusion pump at a constant flow rate every 8 h; (ii) infusion of 0.5 g of doripenem for 1 h via an infusion pump at a constant flow rate every 8 h.

Twelve patients will be enrolled in this study. After completion of the doripenem therapy for 3 days in this study, all patients will receive other sensitive antibiotics to eradicate their bacterial infections.

Sample collections:

Doripenem pharmacokinetic study will be carried out during the doripenem therapy.

Blood samples (approximately 2 ml) in group " 0.5 g of doripenem with 4 h infusion every 8 h regimen" will be obtained by direct venepuncture at the following time: 0, 0.5, 1, 2, 3, 4, 4.5, 5, 6, 7 and 8 h after 7th dose of doripenem.

Blood samples (approximately 2 ml) in group " 0.5 g of doripenem with 1 h infusion every 8 h regimen" will be obtained by direct venepuncture at the following time: 1, 1.5, 2, 4, 5, 6, 7 and 8 h after 7th dose of doripenem.

All blood samples will be allowed to clot and then cebtrifuged at 2,000g.

The serum obtained will be stored at-80°C until analysis.

Doripenem assay:

The doripenem assays by method of Ikeda K et al. (J Chromatogr B, 2008) will be performed at Department of Medicine, Faculty of Medicine.

Clinical data and pathogens collection:

1. Initial patient demographic data (age, sex, weight, diagnosis, APACHE II scores) will be collected upon enrollment in the study.
2. The Gram negative bacilli isolated from sputum in 12 patients will be collected and the MIC of the doripenem for pathogens will be determined by E tests upon enrollment in the study.

Duration of study:

Patients will receive doripenem for 3 days

Pharmacokinetic and pharmacodynamic analysis:

Concentration of doripenem in plasma will be simulated in Monte Carlo technique (Computer model) to get PK/PD index (40%T>MIC) and reported to % PTA (Probability Target Attainment) and %CFR (Cumulative Faction Response)

Sample Size: Twelve patients with VAP will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 20 years
* Patients who have VAP with Gram negative bacilli infections. The diagnosis of VAP was defined by a new and persistent infiltrate on chest radiography associated with at least one of the following: purulent tracheal secretions; temperature of 38.3°C or higher; a leukocyte count higher than 10,000/mm3

Exclusion Criteria:

* Patients who have documented hypersensitivity to doripenem or other carbapenems.
* Patients who have an estimated creatinine clearance of ≤ 50 ml/min
* Patients who are in circulatory shock (defined as a systolic blood pressure of < 90 mmHg).
* Patients who are pregnant.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Concentration of doripenem in plasma | 8 hours profile after 7th dose of doripenem
  Concentration of doripenem in plasma will be simulated in Monte Carlo technique (Computer model) to get PK/PD index (40%T>MIC) and reported to % PTA (Probability Target Attainment) and %CFR (Cumulative Faction Response).

CONTACTS AND LOCATIONS:
Overall Officials: Sutep Jaruratanasirikul, MD, Principal Investigator — Prince of Songkha
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand